CLINICAL TRIAL: NCT02572999
Title: Incidence and Risk Factors for Hospitalization-Associated Disability (HAD) and Its Association With Hospital and Care Processes in Patients With Valvular Heart Disease
Brief Title: Incidence and Risk Factors for Hospitalization-Associated Disability
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: C22/15/028/01
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Functional Decline; Hospitalization-associated Disability; Iatrogenic Disease
Keywords: Aged; Frail; Functional decline; Impairment; valvular heart disease; Cohort; risk factors
MeSH Terms: conditions — Iatrogenic Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Valvular heart disease: All patients aged 70 years or older, consecutively admitted for elective heart valve surgery or if admitted for elective transcatheter aortic valve implantation, or if a patient presents with symptomatic moderate to severe valvular heart disease on hospital admission as evidenced by moderate to severe valve regurgitation or stenosis will be included in this cohort. Participants will be observed up to 30 days post-hospital discharge
  Interventions: Procedure: Not applicable (observational design)

INTERVENTIONS:
Procedure: Not applicable (observational design)

SUMMARY:
This prospective cohort study aims to determine the incidence of hospitalization-associated disability and its association with risk factors at the patient level and with care and hospital processes. For this, patients aged 70 years or older admitted for elective valve surgery or elective transcatheter aortic valve implantation or as a result of symptomatic moderate to severe valvular heart disease will be consecutively included from 01 October 2015 to 29 February 2016.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Admitted for elective heart valve surgery (replacement, repair or combined with CABG) or if admitted for elective transcatheter aortic valve implantation, or if a patient presents with symptomatic moderate to severe valvular heart disease on hospital admission as evidenced by moderate to severe valve regurgitation (≥ 2/4) or aortic valve area ≤ 1cm2 or mitral valve area ≤ 1.5cm2 and if one of the following symptoms is present: heart failure, decreased exercise tolerance, (exertional) dyspnea, (exertional) angina, (exertional) syncope
* Dutch speaking

Exclusion Criteria:

* Life expectancy less than 6 months
* Expected length of stay less than 48 hours

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 70 years and older admitted for elective heart valve surgery (replacement, repair or combined with CABG) or if admitted for elective transcatheter aortic valve implantation, or if a patient presents with symptomatic moderate to severe valvular heart disease on hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hospitalization-associated Disability | Up to 30 days post-hospital discharge
  The loss of ability to complete one of the basic ADLs independently between baseline and hospital discharge.

SECONDARY OUTCOMES:
The six minutes walking distance test | Up to 30 days post-hospital discharge
Five meter gait speed test | Up to 30 days post-hospital discharge
Timed get-up and go test | Up to 30 days post-hospital discharge
Peak extension torque measured at the right side and evaluated at 60° of knee flexion | Up to 30 days post-hospital discharge
  Isometric quadriceps strength will be measured using a dynamometer (Biodex system 4 pro; Enraf Nonius; Delft, The Netherlands)
Peak handgrip force assessed at the dominant side with the elbow at 90° of flexion, and the forearm and wrist in a neutral position. | Up to 30 days post-hospital discharge
  Isometric handgrip force will be measured with a hydraulic hand dynamometer (Jamar dynamometer; JA Preston Corporation; Jackson, MI)
Inappropriate medication prescribing | Up to 30 days post-hospital discharge
  Inappropriate medication prescribing using the RASP-list (Rationalization of Home Medication by an Adjusted STOPP list in Older Patients)

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Deschodt, PhD, Principal Investigator — KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Jonckers M, Van Grootven B, Willemyns E, Hornikx M, Jeuris A, Dubois C, Herregods MC, Deschodt M. Hospitalization-associated disability in older adults with valvular heart disease: incidence, risk factors and its association with care processes. Acta Cardiol. 2018 Jan 4;73(6):566-572. doi: 10.1080/00015385.2017.1421300. PMID 29301463